CLINICAL TRIAL: NCT06744647
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Evaluate Efficacy and Safety of ALXN2030 in Adult Patients With Antibody-Mediated Rejection After Kidney Transplantation
Brief Title: Phase 2 Study of ALXN2030 in Patients With Antibody-Mediated Rejection After Kidney Transplantation
Acronym: CONCORD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8560C00002
Record Dates: First submitted 2024-12-13; First posted 2024-12-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Antibody-Mediated Rejection; Kidney Transplantation; Biopsy-proven Histologic Scores; AMR
Keywords: ALXN2030; Antibody-Mediated Rejection; Kidney Transplantation; Biopsy-proven histologic scores; AMR

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo will be administered during the Double-Blind Treatment Period of 52 weeks.
  Interventions: Drug: Placebo
- ALXN2030 Dose A (Experimental): During the Double-Blind Treatment Period, participants will receive ALXN2030 dose A over 52 weeks. At Week 52, participants may continue into the Open Label Extension (OLE).
  Interventions: Drug: ALXN2030
- ALXN2030 Dose B (Experimental): During the Double-Blind Treatment Period, participants will receive ALXN2030 dose B over 52 weeks. At Week 52, participants may continue into the OLE Period.
  Interventions: Drug: ALXN2030

INTERVENTIONS:
Drug: ALXN2030 — ALXN2030 will be administered subcutaneously (SC).
  Arms: ALXN2030 Dose A; ALXN2030 Dose B
Drug: Placebo — Placebo will be administered SC.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of ALXN2030 compared with placebo on biopsy proven histologic resolution in participants with active or chronic active antibody-mediated rejection (AMR) at Week 52.

DETAILED DESCRIPTION:
This prospective trial will assess the efficacy, safety, pharmacokinetics, pharmacodynamics, and immunogenicity of ALXN2030 in kidney transplant recipients with active or chronic active AMR. The study is designed as a randomized, controlled, double-blind phase 2 trial. Participants will be randomized in a 1:1:1 ratio to receive either ALXN2030 Dose A, ALXN2030 Dose B, or placebo for a double-blind treatment period of 52 weeks. All arms will receive standard of care immunosuppressive treatment. During the treatment period, study participants will be subjected to repeated allograft biopsies at 28 and 52 weeks. At the end of the double-blind treatment period, participants may continue into the Open-Label Extension (OLE) Treatment Period (52 weeks). Participants randomized to placebo will be re-randomized 1:1 to ALXN2030 Dose A or ALXN2030 Dose B. Safety Follow-Up will start after the end of Treatment (Week 104) until week 48 after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant received ≥ 6 months
* Active or chronic active AMR according to Banff 2022 classification, based on Screening kidney biopsy
* Either positive C4d on Screening kidney biopsy based on the Central Pathology Laboratory report and/or positive HLA Class I and/or II antigen-specific DSA as determined by the local laboratory's definition of positivity using single-antigen bead based assays
* MVI score ≥ 2 (g ≥ 1 and ptc ≥ 1)
* eGFR ≥ 30 mL/min/1.73 m2
* Must be vaccinated against meningococcal infection from serogroups A, C, W, Y (and B where available) at least 14 days prior to but no more than 3 years prior to Day 1
* Must be vaccinated for S pneumoniae prior to randomization
* Must be vaccinated for H influenzae type B (where available) prior to randomization
* Body weight ≥ 50 kg at Screening

Exclusion Criteria:

* Biopsy-based diagnosis of any of the following at Screening:
* TCMR, according to the Banff grade ≥ 1
* Polyoma virus nephropathy
* Severe thrombotic microangiopathy
* Glomerulonephritis
* ABO-incompatible transplant
* uACR > 2200 mg/g
* Multiorgan transplant recipient (except for previous multiple kidney transplants) or cell transplant (islet, bone marrow, stem cell) recipient
* Planned or recent treatments, < 3 months prior to the Screening Visit, for Acute Rejection, AMR (including plasmapheresis, plasma exchange, IVIg, B-cell depleting therapy, IL inhibitors, proteasome inhibitors, high-dose corticosteroids [except for tapering]), TCMR (including T-cell depleting therapy), excluding the SoC immunosuppressant treatment which will be allowed and should be stable during the entire treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2027-10-11 (Estimated); Study Completion 2028-11-07 (Estimated)

PRIMARY OUTCOMES:
Biopsy-proven histologic resolution | Week 52

SECONDARY OUTCOMES:
Biopsy-proven histologic resolution | Week 28
Change From Baseline in biopsy-proven histologic scores | Baseline, Weeks 28 and 52
Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 52 | Baseline up to week 52
Annualized Total eGFR Slope | Baseline up to Week 52
Stabilized eGFR | Baseline up to Week 52
Number of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (TESAEs) | Day 1 up to Week 104
Number of Participants With Anti-drug Antibodies (ADAs) | Day 1 through Week 104
Plasma Concentration of ALXN2030 | Baseline up to Week 104
Plasma Concentration of C3 Protein | Baseline up to Week 104
Change From Baseline in Serum Complement Functional Activity | Baseline, up to Week 52 and up to Week 104

CONTACTS AND LOCATIONS:
Locations (44):
- United States (20):
  - Research Site, Birmingham, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Kansas City, Kansas
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Livingston, New Jersey
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin
- Brazil (4):
  - Research Site, Botucatu
  - Research Site, Campinas
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Canada (6):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (6):
  - Research Site, Changsha
  - Research Site, Guangzhou
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Wuhan
  - Research Site, Xi'an
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Zaragoza
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taoyuan District
- United Kingdom (2):
  - Research Site, Birmingham
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR